CLINICAL TRIAL: NCT04495205
Title: Clinical Comparison of the Effect of Non-eugenol Containing Periodontal Pack With and Without Platelet Rich Fibrin on Post-operative Pain and Wound Healing After Surgical Gingival Depigmentation: A Randomized Clinical Trial
Brief Title: Effect of Non-eugenol Periodontal Pack With and Without PRF on Post-operative Pain and Wound Healing After Gingival Depigmentation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Hesham Reda, Masters Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AHReda
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Gingival Pigmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the statistician are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-eugenol containing periodontal packs with PRF (Experimental): Non-eugenol containing periodontal packs with PRF after gingival de-pigmentation
  Interventions: Biological: PRF under non-eugenol containing periodontal pack
- Non-eugenol containing periodontal packs (Placebo Comparator): Non-eugenol containing periodontal packs after gingival de-pigmentation
  Interventions: Other: Non-eugenol containing periodontal pack

INTERVENTIONS:
Biological: PRF under non-eugenol containing periodontal pack — Platelet Rich Fibrin under non-eugenol containing periodontal pack
  Other Names: Platelet Rich Fibrin
  Arms: Non-eugenol containing periodontal packs with PRF
Other: Non-eugenol containing periodontal pack — Non-eugenol containing periodontal pack after gingival depigmentation
  Arms: Non-eugenol containing periodontal packs

SUMMARY:
In an era where less than ideal esthetics is not accepted, the request for esthetic procedures is widely sought after. Melanin, a brown pigment, is the most common natural pigment contributing to endogenous pigmentation of gingiva. It is a non-hemoglobin-derived pigment formed by cells called melaonocytes

Dental cosmetic procedures including gingival depigmentation among the young generation are vastly becoming popular due to the public advertising of what the "ideal smile" should be. This means that brown/ pigmented gingiva is not esthetically accepted by modern standards. Numerous techniques for depigmentation were developed including surgical abrasion, lasers, chemicals and thermal techniques.

The use of post-operative non-eugenol containing periodontal packs acts as a mechanical barrier for coverage of the denuded area which prevents bleeding and promotes healing by preventing trauma to the area.

Platelet Rich Fibrin (PRF) is a form of concentrated suspension of growth factors that promote healing and tissue regeneration. Its use in the medical and dental fields is expanding during the recent year.

DETAILED DESCRIPTION:
Gingival depigmentation procedures especially bur abrasion and scalpel surgical techniques require the use of post-operative periodontal pack. The periodontal pack protects the surgical site from surface trauma, stops the post-operative bleeding and infection as well as stabilizing the blood clot and accelerate healing.

However, a review article discussed the adverse effects of periodontal pack as it may cause plaque induced inflammation, patient discomfort due to difficulty in eating and irritation of the tissues. In the article, there were clinical trials that advocated that wound healing could occur without the need of periodontal pack if the surgical wound was kept clean alone indicating that the pack does not affect the wound healing.

This gave rise to idea to use a material that has been proven to accelerate wound healing and decrease the patient discomfort to be placed under the periodontal pack which would be used only as a protective barrier.

Several studies tested platelet rich concentrates as adjunctive methods under periodontal packs verses periodontal packs alone after surgical abrasion of gingival depigmentation. They found that there was a clinical, histological and statistical difference between the groups favoring the platelet concentrate groups.

Using PRF which is a second generation platelet concentrate first developed by Choukroun et al in 2001 used as a membrane could provide accelerated wound healing properties which would accelerate ginigival re-epithelization . Using a periodontal pack is conventionally used which will provide a mechanical barrier to protect the wound from any stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Ages18-40 years old
* Systemically healthy
* Mild to moderate gingival pigmentations
* Gingival and plaque index <1
* Good oral hygiene
* Thick gingival biotypes
* Keratinized gingiva >2mm

Exclusion Criteria:

* Smokers
* Taking any medications that could affect healing
* Pervious depigmentation procedures
* Pregnant or lactating females
* Pervious periodontal surgery within the last 6 months before the start of the trial
* Endodontically treated teeth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 1st day post-operative
  Visual Analog Scale: minimum score 0 (no pain), maximum score 10 (unbearable pain)
Post-operative pain | 3rd day post-operative
  Visual Analog Scale: minimum score 0 (no pain), maximum score 10 (unbearable pain)
Post-operative pain | 5th day post-operative
  Visual Analog Scale: minimum score 0 (no pain), maximum score 10 (unbearable pain)

SECONDARY OUTCOMES:
Re-epithelization | 5th day post-operative
  Toulodine Blue test: dark blue = positive (worst score), light blue = negative (better score)
Wound healing | 3rd day post-operative
  Healing Index (Landry, 1985): minimum score 1 (very poor), maximum score 5 (excellent)
Wound healing | 5th day post-operative
  Healing Index (Landry, 1985): minimum score 1 (very poor), maximum score 5 (excellent)
Re-pigmentation | 6 months post-operative
  Re-pigmentation of de pigmented site (Kumar, Bhat and Bhat, 2012): minimum score 0 (absence of depigmentation, maximum score 3 (Diffuse brown to black pigmentation, marginal, and attached)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahiya R, Blaggana A, Panwar V, Kumar S, Kathuria A, Malik S. Clinical and histological comparison of platelet-rich fibrin versus non-eugenol periodontal dressing in the treatment of gingival hyperpigmentation. J Indian Soc Periodontol. 2019 Jul-Aug;23(4):345-350. doi: 10.4103/jisp.jisp_688_18. PMID 31367132